CLINICAL TRIAL: NCT03112369
Title: Preventing HIV Among Native Americans Through the Treatment PTSD & Substance Use
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Cynthia Pearson, Professor, Director of Research, Indigenous Wellness Research Institute School of Social Work, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: STUDY00001359; R01MD011574 (NIH)
Record Dates: First submitted 2017-04-10; First posted 2017-04-13 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: HIV Prevention; PTSD and Substance Use Disorder
Keywords: American Indian / Alaska Native; HIV Prevention; Sexual Risk Behavior; Trauma; Substance Use
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Substance-Related Disorders; Wounds and Injuries

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Narrative Exposure Therapy (NET) (Experimental): Counseling program
  Interventions: Behavioral: Narrative Exposure Therapy (NET)
- Motivational Interviewing w/Skills Training (MIST) (Experimental): Counseling program
  Interventions: Behavioral: Motivational Interviewing w/Skills Training (MIST)

INTERVENTIONS:
Behavioral: Narrative Exposure Therapy (NET) — An international evidence-based program (EBP) for PTSD based on exposure therapy, an oral tradition of story-telling, and use of tactile medium of natural elements.
  Arms: Narrative Exposure Therapy (NET)
Behavioral: Motivational Interviewing w/Skills Training (MIST) — Motivational interviewing (MI) coupled with skills training is based on enhancing motivation to change and building skills to address substance use behaviors.
  Arms: Motivational Interviewing w/Skills Training (MIST)

SUMMARY:
Investigators will conduct a two-arm, comparative effectiveness randomized controlled trial of two culturally adapted, empirically based programs (EBP) - Narrative Exposure Therapy (NET) vs. Motivational Interviewing with Skills Training (MIST) in terms of lowering HIV sexual-risk behaviors (HSB) for American Indian / Alaska Native (AIAN) men and women. NET addresses Posttraumatic Stress Disorder (PTSD) as a pathway to preventing substance use disorders (SUD) and HSB whereas MIST addresses substance misuse as a way of preventing SUD and HSB.

DETAILED DESCRIPTION:
Recruitment Participants will be recruited from tribal health and wellness service agencies and counseling centers on the Reservation as well as through advertising in the community. Investigators will post flyers in public spaces like coffee shops, the library, the cultural center, and community centers. We will also send the flyer through the tribal listserv; post it on Facebook, and the local newspaper. Investigators will provide brief oral presentations at the local health centers to orient providers of the project and provide contact information and flyers. Providers and potential participants who are interested may contact the study coordinator for more information

Screening

* Participants are screened in person or over the phone using a screening script.
* Participants who screen out will be given a community resource list either by mail, email, or in person.
* If a person is eligible but declines to participate, they will be given a one item exit question regarding general reason for non-participation.

Consent and Baseline Assessment After completing the screener, the participant will be scheduled for an in-person consenting / baseline assessment appointment. Study staff will review the consent form with the participant. Once participant has consented, study staff will gather all relevant contact information. Next, study staff will set up the computer for the participant to complete the Audio Computer Assisted Self-interview (ACASI) survey, which will take approximately 30 minutes. While the participant is completing the survey, local study staff will call the Research Coordinator (RC) to confirm the consent has been obtained and to determine randomization. The RC will let the local study staff know which counselor the person should be scheduled with for the 1st counseling appointment. The counselor will inform which therapy the participant was assigned to at their first counseling session. Once participant completes the computer survey, study staff will schedule their first counseling appointment to take place within a week of the baseline appointment.

Assessments The assessments will be conducted via Audio-Computer Assisted Self-Interviews (ACASI) programmed into study computers. Participants will complete 4 surveys: baseline, immediately after completing counseling, a three-month follow up and a six-month follow up.

Counseling sessions Participants will be randomly assigned to either NET or MIST. To ensure the equivalence of groups and to reduce opportunities for selection bias we will stratify the randomization by gender (male vs. female) and age groups (<30 vs. >=30) and perform randomization in blocks with varying size (4/6/8). Participants will begin their six 90 to 120 minute sessions in within a week of completing the Baseline assessment. Each counseling session is audio recorded in order for investigators to test for fidelity and adherence to the culturally adapted therapy.

ELIGIBILITY:
Inclusion Criteria:

* 16 years old or older
* Native American
* At least sub-threshold PTSD
* Substance use in the previous 12 months
* Any lifetime sexual activity

Exclusion Criteria:

* Suicidal ideation, plan, or attempt in the previous 30 days
* Homicidal ideation in the previous 3 months
* Psychiatric medication that has not been stable for at least 2 months
* A DSM-5 alcohol dependence diagnosis with severe withdrawal symptoms

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2017-09-21 (Actual); Primary Completion 2024-08-16 (Actual); Study Completion 2024-08-30 (Actual)

PRIMARY OUTCOMES:
National Institute on Drug Abuse (NIDA) Seek, Test, Treat and Retain for Vulnerable Populations: Data Harmonization Measure | Baseline and Post Intervention; Baseline and 3-month Follow up; Baseline and 6-month Follow up
  Measuring change in high risk sexual behavior for contracting HIV.
Change in Drug Use as assessed by PhenX Toolkit | Baseline and Post Intervention; Baseline and 3-month Follow up; Baseline and 6-month Follow up
  This measure is used to assess changes in participant's substance use.
Change in PTSD symptoms as assessed by the Posttraumatic Symptom Scale Interview Diagnostic and Statistical Manual 5th Ed (DSM-5) (PSSI5) | Baseline and Post Intervention; Baseline and 3-month Follow up; Baseline and 6-month Follow up
  This measure is used to assess the severity of the PTSD symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia R Pearson, PhD, Principal Investigator — University of Washington; Debra Kaysen, PhD, Principal Investigator — Stanford University
Locations (1):
- University of Washington School of Social Work, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: Yes
Only De-identified IPD will be available after institutional IRB and tribal approval

REFERENCES:
- [Background] Walker D, Pearson C, Day A, Bedard-Gilligan M, Saluskin K, Huh D, Kaysen D. A Community Engaged Approach in Adapting Motivational Interviewing and Skills Training for Native Americans With Experiences of Substance Misuse. Am J Health Promot. 2023 Jul;37(6):796-806. doi: 10.1177/08901171231161467. Epub 2023 Mar 4. PMID 36869715
- [Background] Bedard-Gilligan M, Kaysen D, Cordero RM, Huh D, Walker D, Kaiser-Schauer E, Robjant K, Saluskin K, Pearson C. Adapting narrative exposure therapy with a tribal community: A community-based approach. J Clin Psychol. 2022 Nov;78(11):2087-2108. doi: 10.1002/jclp.23395. Epub 2022 May 27. PMID 35621371
- [Background] Pearson CR, Kaysen D, Huh D, Bedard-Gillgan M, Walker D, Marin R, Saluskin K. A randomized comparison trial of culturally adapted HIV prevention approaches for Native Americans reducing trauma symptoms versus substance misuse: The Healing Seasons protocol. Contemp Clin Trials. 2020 Aug;95:106070. doi: 10.1016/j.cct.2020.106070. Epub 2020 Jun 17. PMID 32561467